CLINICAL TRIAL: NCT04796415
Title: Daily Engagement in Meaningful Activities Professional (DEMA-Pro) Intervention for Seniors With Subjective Cognitive Decline and Living at Home
Brief Title: DEMA-Pro Intervention for Seniors With Subjective Cognitive Decline and Living at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Yvonne Lu, Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 00622607; R61 AG07265-01 (Other Grant/Funding Number: NIA)
Record Dates: First submitted 2021-02-03; First posted 2021-03-12 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Subjective Cognitive Decline
Keywords: DEMA-Pro; daily meaningful activity; cognitive impairment; caregivers
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DEMA-Pro (Experimental): The DEMA-Pro intervention will be administrated. Subjects will attend six weekly, 1-hour telephone sessions.
  Interventions: Behavioral: the DEMA-Pro intervention

INTERVENTIONS:
Behavioral: the DEMA-Pro intervention — Trained DEMA-Pro coaches will deliver six weekly, 1-hour telephone sessions. The first session is an orientation to the DEMA-Pro intervention and development of the initial Weekly Activity Plan based on the patient's self-identified meaningful activity. Over the next five weekly sessions, the coach uses problem-solving strategies to facilitate dyad collaboration to mutually identify meaningful activities and make a realist plan to achieve the patient-identified meaning activity goals. In each session, the patient and caregiver also select, review, and discuss one of six topics in the Self-Management Toolkit (e.g., planning meaningful activities; learning strategies for living with subjective cognitive impairment; finding resources, planning for the future).

SUMMARY:
More than 4.4 million patients receive home health services following discharge from the hospital or rehabilitation facility. A substantial number (70%) are older adults with subjective cognitive decline (SCD), an early clinical sign of Alzheimer's disease and related dementia. SCD is associated with diminished activity performance, poor quality-of-life and other adverse health outcomes (e.g., depressive symptoms). Home health patients with SCD often require more time, structure, and guidance to complete tasks and adjust to new skills and environments. Support is especially important during this high-risk period of transition between care settings. We propose a new home health care delivery model in partnership with Kindred at Home (KAH), a division of Humana that encompasses 400 programs across 40 states. DEMA-Pro builds on five preliminary studies that demonstrated high feasibility, acceptability, and positive preliminary effects on health outcomes (physical function, mood, and QoL). DEMA-Pro will be refined for delivery by home health services staff to patients with SCD and their informal caregivers. The overall goal of this research will be to conduct a pragmatic cluster randomized controlled trial (RCT) of DEMA-Pro to improve outcomes in-home health service patients with SCD. In the current R61 pilot phase, we will establish the trial's organizational structure and processes and pilot test DEMA-Pro in 4 home health services sites. In a subsequent trial, we plan to conduct a full pragmatic RCT in a group of Kindred KAH sites comparing DEMA-Pro to usual care. Consistent with the spirit of a pragmatic trial, we will use existing data sources including electronic Medicare OASIS (Outcome and Assessment Information Set) data, and QoL to characterize the cohort and measure outcomes. Thus, the focus of the pilot phase will be to ensure all processes are in place to conduct the subsequent RCT.

Aim 1. Establish the organizational infrastructure and programmatic processes needed to conduct a pragmatic cluster-randomized control trial of the DEMA-Pro intervention versus usual care. A Steering Committee will lead the project and coordinate the activities of 3 Work Groups: Regulatory and Operations; DEMA-Pro Intervention Protocol; and Data Management and Analysis.

Aim 2. Pilot test the DEMA-Pro training protocol in 4 KAH North Region locations and refine as indicated.

ELIGIBILITY:
Inclusion Criteria for Home Health patients

* 1) Home health service patients aged > 50 years with SCD, with an OASIS- Cognition Function Subscale Score of 1 or 2 (0 = alert/oriented, able to focus and shift attention, comprehends and recalls task directions independently; 1 = Requires prompting [cuing, repetition, reminders) only under stressful or unfamiliar conditions; 2 = Requires assistance and some direction in specific situations [for example, on all tasks involving shifting of attention] or consistently requires low stimulus environment due to distractibility; 3 = Requires considerable assistance in routine situations. Is not alert and oriented or is unable to shift attention and recall directions more than half the time; 4 = Totally dependent due to disturbances such as constant disorientation, coma, persistent vegetative state, or delirium.

Exclusion:

-No caregiver

Criteria for home health services sites are: 1) a minimum of 300 or more new patients/per site annually; 2) at least 50% w/ length of service > 60 days; 3) staff-to-patient ratio complies with Home Health Agency requirements; 4) no severe state issues. Prior to randomization, sites meeting these criteria will be determined in consultation with the KAH, Clinical Operations Coordinator.

* KAH staff including call-center care coordinators, clinical assessment associates, field-based therapists, and clinical operational coordinator

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Lu, PhD, RN, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Kindred at Home, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patient enrollment is reported because patients were the pre-specified participants. Feedback about the intervention was collected from staff, but staff were not participants.
Period: Overall Study
Arm/Group | DEMA-Pro
Started (Completed OASIS at starting date; eligible Home Health Care patients and initial Call) | 49
Session #1 | 35
Session #2 | 25
Session #3 | 21
Session #4 | 19
Session #5 | 19
Session #6 | 18
Completed | 18
Not Completed | 31
Not completed — not interested | 12
Not completed — health issue | 8
Not completed — Other | 4
Not completed — discharged from home health service | 3
Not completed — re-hospitalization | 2
Not completed — moving to nursing home | 1
Not completed — lost contact | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics for patients are included. No baseline characteristics were collected from staff because they were not pre-specified participants
Arm/Group | DEMA-Pro
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 44
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean Age | 78.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 44
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 49
Primary Diagnosis [Count of Participants; unit: Participants]
  Diabetes | 21
  Cardiovascular related | 33
  Primary Diagnosis related to fracture, surgery and post-surgery care | 16
  Participants with hospitalization risks | 49

OUTCOME MEASURES:

1. Primary Outcome: Physical Function
Description: Change in Physical Function measured by the Outcome and Assessment Information Set Data of Instructive Activities of Daily Living Scale (OASIS-D, IADLs Scale M1800s ).The ADL/IADL composite score ranges from 0 (total independence) to 9 (totally dependent/unable to complete). Higher score represent greater dependence.
Time Frame: Baseline to 6 weeks
Population: 14/18 completed OASIS-D ADLs Scale at start of care (pre- intervention) and when discharged from Home Health Agency(post-intervention) in this Pilot Phase of pragmatic trial.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- DEMA-Pro: The DEMA-Pro intervention will be administered. Subjects will attend six weekly, 1-hour telephone sessions.
  the DEMA-Pro intervention: Trained DEMA-Pro coaches will deliver six weekly, 1-hour telephone sessions. The first session is an orientation to the DEMA-Pro intervention and development of the initial Weekly Activity Plan based on the patient's self-identified meaningful activity. Over the next five weekly sessions, the coach uses problem-solving strategies to facilitate dyad collaboration to mutually identify meaningful activities and make a realist plan to achieve the patient-identified meaning activity goals. In each session, the patient and caregiver also select, review, and discuss one of six topics in the Self-Management Toolkit (e.g., planning meaningful activities; learning strategies for living with subjective cognitive impairment; finding resources, planning for the future).
Arm/Group | DEMA-Pro
Number analyzed (Participants) | 14
score on a scale | -4.7 (1.2)

2. Secondary Outcome: Sense of Well-Being
Description: Psychosocial Well-being-Short-Form.The Psychosocial well-being short form composes 12 items and ranges from 12 to 60. Higher scores represent better quality of life.Change in the mean score and standard deviation was calculated from pre and post DEMA-Pro intervention. 1-5 Likert Scale. 1= not at all, 5= very much or strongly agree
Time Frame: 1 week before DEMA-Pro intervention and post-DEMA-Pro program within 10 days
Population: 18 participants psychosocial well-being measures was collected by Home Health Agency Call Center Staff at pre and post DEMA-Pro program..
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DEMA-Pro
Number analyzed (Participants) | 18
score on a scale | 7.7 (4.6)

3. Secondary Outcome: Depression
Description: OASIS-D sub data of PHQ-2 (M1730); The current version of OASIS does not have PhQ-2 items so we did not ask the coach to collect the PHQ-2 data.
Time Frame: 1 week before DEMA-Pro intervention and post-DEMA-Pro program within 10 days
Population: The OASIS PHQ-2 was not collected because the current version of OASIS-D does not have PHQ-2 subscale.
Arm/Group | DEMA-Pro
Number analyzed (Participants) | 0

4. Secondary Outcome: Hospitalization Rate
Description: OASIS-D sub data of Frequency of rehospitalization rate (M2410)
Time Frame: One year after completing the intervention
Population: Outcome data collection was not funded for this measure, data were not collected
Arm/Group | DEMA-Pro
Number analyzed (Participants) | 0

5. Secondary Outcome: Number, Types of ER Visits
Description: OASIS-D sub data of Frequency unplanned urgent care or hospital ER care (M2301, M2041)
Time Frame: One year after completing the intervention
Population: Outcome data collection was not funded for this measure, so data were not collected.
Arm/Group | DEMA-Pro
Number analyzed (Participants) | 0

6. Secondary Outcome: Nursing Home Transfers
Description: OASIS-D sub data of Frequency of transfers to nursing home care (M2410)
Time Frame: One year after intervention
Population: .Outcome data collection was not funded for this measure, so data were not collected.
Arm/Group | DEMA-Pro
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year 3 months
Description: Adverse events for patients, who were the pre-specified participants, are included. Adverse events were not collected or reported for staff.
Arm/Group | DEMA-Pro
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 4/49
Other Adverse Events (participants affected / at risk) | 3/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DEMA-Pro (N=49)
Visited ED due to fall and fracture of 2 ribs (Vascular disorders) | 1 (1) — fractured 2 ribs without hospitalization
Hospitalization (Cardiac disorders) | 1 (1) — due to low blood pressure
Visited ED due to high blood pressure 228/119 (Vascular disorders) | 1 (1)
Hospitalization due to CHF (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DEMA-Pro (N=49)
Fall without injury (General disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Small sample sizes, potential bias due lack of discharge/transfer outcome being collected, lack of true control group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/15/NCT04796415/Prot_SAP_000.pdf